CLINICAL TRIAL: NCT06239103
Title: Effectiveness of Pulsed Electromagnetic Field Therapy as an Adjunct Modality to Warm-up Exercise: a Randomized Controlled Trial
Brief Title: Effect of Pulsed Electromagnetic Field Therapy as an Adjunct Modality to Warm-up Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Justine Tin Nok Chan, Medical Student Researcher, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 202.616-T
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Knee Range-of-motion; Quadriceps Muscle Stiffness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEMF treatment arm (Experimental): Participants receive PEMF therapy. During this, the participant is seated with their right leg extended and with the bore of the PEMF machine between their knee and hip joints, with their left leg at rest. PEMF was applied at 1 mT, 15 Hz for 10 minutes.
  Interventions: Device: Pulsed electromagnetic field therapy
- Control arm (Sham Comparator): Participants receive sham therapy, where the PEMF machine does not apply the pulsed electromagnetic waves. However, during this, the participant is kept in the same position as those in the treatment arm.
  Interventions: Device: Sham treatment

INTERVENTIONS:
Device: Pulsed electromagnetic field therapy — Pulsed electromagnetic field therapy for 10 minutes, using a PEMF device, at 1 mT, 15 Hz.
  Arms: PEMF treatment arm
Device: Sham treatment — Sham treatment, using the same PEMF device
  Arms: Control arm

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of pulsed electromagnetic field therapy as an adjunct to warm-up exercises, in healthy participants. Researchers will investigate both the immediate effect of one round of pulsed electromagnetic field therapy (PEMF) and after a warm-up exercise, on participants' range-of-motion (ROM) at the knee and quadriceps' muscle stiffness, measured through shear wave elastography, an ultrasound technique. This may be useful in future interventions to protect against sports injuries.

Participants will have their knee ROM and quadriceps' muscle stiffness measured thrice, once at baseline, once after PEMF/sham treatment, and once after 5 minutes of warm-up stationary bike exercises.

Researchers will compare with sham treatment to see if there are any significant effects from PEMF therapy.

DETAILED DESCRIPTION:
The goal of this clinical trial is to assess the effectiveness of pulsed electromagnetic field therapy as an adjunct to warm-up exercises, in healthy participants. Researchers will investigate both the immediate effect of one round of pulsed electromagnetic field therapy (PEMF) and after a warm-up exercise, on participants' range-of-motion (ROM) at the knee and quadriceps' muscle stiffness, measured through shear wave elastography, an ultrasound technique. This may be useful in future interventions to protect against sports injuries.

Participants will have their knee ROM and quadriceps' muscle stiffness measured thrice, once at baseline, once after PEMF/sham treatment, and once after 5 minutes of warm-up stationary bike exercises.

* Baseline measurement of knee ROM and quadriceps' muscle stiffness
* Receive PEMF for ten minutes around their knee joint
* Interim measurement of knee ROM and quadriceps' muscle stiffness
* Perform 5 minutes of warm-up exercise on a stationary bike
* Final measurement of knee ROM and quadriceps' muscle stiffness

Researchers will compare with sham treatment to see if there are any significant effects from PEMF therapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40
* Obtained written informed consent

Exclusion Criteria:

* History of major musculoskeletal or locomotor system disorder of lower limb
* History of traumatic or non-traumatic injury of lower limb
* History of surgical intervention of lower limb in the past 1 year
* Under any rehabilitation program at the time of investigation
* Contraindicated to physical exercises

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Change in knee range-of-motion from baseline immediately after PEMF and after warm-up exercise, as assessed by goniometer | From before PEMF/sham treatment to end of treatment and warm-up exercise, within 1 hour
  A goniometer will be used to measure the knee range-of-motion: the static arm will follow a line joining the knee to the greater trochanter of the femur, and the moving arm a line from the knee to the lateral malleolus of the ankle

SECONDARY OUTCOMES:
Change in quadriceps muscle stiffness from baseline immediately after PEMF and after warm-up exercise, as assessed by ultrasound shear wave elastography | From before PEMF/sham treatment to end of treatment and warm-up exercise, within 1 hour
  Ultrasound imaging and shear wave elastography will be used to measure the stiffness of the three superficial quadriceps muscles (vastus medialis, vastus lateralis and rectus femoris). Markings will be made to standardise the position of scanning. Ultrasound imaging will be used to verify the muscle being scanned. After shear wave is applied and a stable image is obtained, Young's modulus will be measured as a measure of muscle stiffness.

CONTACTS AND LOCATIONS:
Overall Officials: Justine Tin Nok Chan, Principal Investigator — University of Cambridge
Locations (1):
- CUHK-ORT Sports Injury Research Laboratory, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No